CLINICAL TRIAL: NCT03672188
Title: A Phase 1/2, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of VIR-2218
Brief Title: Study of VIR-2218 in Healthy Subjects and Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Collaborators: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIR-2218-1001
Record Dates: First submitted 2018-09-11; First posted 2018-09-14 (Actual); Results first posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B Virus; Chronic Hepatitis B; HBV; Hepatitis
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Hepatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (15):
- Part A: SAD VIR-2218 50 mg (Experimental): Healthy subjects received a single dose of VIR-2218 of 50 mg administered SC
  Interventions: Drug: VIR-2218
- Part A: SAD VIR-2218 100 mg (Experimental): Healthy subjects received a single dose of VIR-2218 of 100 mg administered SC
  Interventions: Drug: VIR-2218
- Part A: SAD VIR-2218 200 mg (Experimental): Healthy subjects received a single dose of VIR-2218 of 200 mg administered SC
  Interventions: Drug: VIR-2218
- Part A: SAD VIR-2218 400 mg (Experimental): Healthy subjects received a single dose of VIR-2218 of 400 mg administered SC
  Interventions: Drug: VIR-2218
- Part A: SAD VIR-2218 600 mg (Experimental): Healthy subjects received a single dose of VIR-2218 of 600 mg administered SC
  Interventions: Drug: VIR-2218
- Part A: SAD VIR-2218 900 mg (Experimental): Healthy subjects received a single dose of VIR-2218 of 900 mg administered SC
  Interventions: Drug: VIR-2218
- Part A: SAD Placebo (Placebo Comparator): Healthy subjects received a single dose of placebo administered SC
  Interventions: Drug: Placebo
- Part B: MAD VIR-2218 20 mg (Experimental): Chronic HBV, HBeAg negative, subjects received 2 SC doses of 20 mg VIR-2218 administered 4 weeks apart.
  Interventions: Drug: VIR-2218
- Part B: MAD VIR-2218 50 mg (Experimental): Chronic HBV, HBeAg negative, subjects received 2 SC doses of 50 mg VIR-2218 administered 4 weeks apart.
  Interventions: Drug: VIR-2218
- Part B: MAD VIR-2218 100 mg (Experimental): Chronic HBV, HBeAg negative, subjects received 2 SC doses of 100 mg VIR-2218 administered 4 weeks apart.
  Interventions: Drug: VIR-2218
- Part B: MAD VIR-2218 200 mg (Experimental): Chronic HBV, HBeAg negative, subjects received 2 SC doses of 200 mg VIR-2218 administered 4 weeks apart.
  Interventions: Drug: VIR-2218
- Part C: MAD VIR-2218 50 mg (Experimental): Chronic HBV, HBeAg positive, subjects received 2 SC doses of 50 mg VIR-2218 administered 4 weeks apart.
  Interventions: Drug: VIR-2218
- Part C: MAD VIR-2218 200 mg (Experimental): Chronic HBV, HBeAg positive, subjects received 2 SC doses of 200 mg VIR-2218 administered 4 weeks apart.
  Interventions: Drug: VIR-2218
- Part B: MAD Placebo (Placebo Comparator): Chronic HBV, HBeAg negative, subjects received 2 SC doses of placebo administered 4 weeks apart.
  Interventions: Drug: Placebo
- Part C: MAD Placebo (Placebo Comparator): Chronic HBV, HBeAg positive, subjects received 2 SC doses of placebo administered 4 weeks apart.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIR-2218 — VIR-2218 given by subcutaneous injection
  Arms: Part A: SAD VIR-2218 100 mg; Part A: SAD VIR-2218 200 mg; Part A: SAD VIR-2218 400 mg; Part A: SAD VIR-2218 50 mg; Part A: SAD VIR-2218 600 mg; Part A: SAD VIR-2218 900 mg; Part B: MAD VIR-2218 100 mg; Part B: MAD VIR-2218 20 mg; Part B: MAD VIR-2218 200 mg; Part B: MAD VIR-2218 50 mg; Part C: MAD VIR-2218 200 mg; Part C: MAD VIR-2218 50 mg
Drug: Placebo — Sterile normal saline (0.9% NaCl) given by subcutaneous injection
  Arms: Part A: SAD Placebo; Part B: MAD Placebo; Part C: MAD Placebo

SUMMARY:
This is a phase 1/2 study in which healthy adult subjects and subjects with chronic hepatitis B virus (HBV) infection will receive VIR-2218 or placebo and will be assessed for safety, tolerability, pharmacokinetics, and antiviral activity (only in subjects with chronic HBV).

In the single ascending dose (SAD) part, Part A, healthy adult subjects will receive one dose of VIR-2218 or placebo, administered subcutaneously (SC). In the multiple ascending dose (MAD) parts, Part B & Part C, subjects with chronic HBV infection will receive two doses of VIR-2218 or placebo every 4 weeks administered SC.

ELIGIBILITY:
Part A SAD:

Inclusion Criteria:

* Male or female age 18 - 55
* BMI 18 - 32 kg/m^2

Exclusion Criteria:

* Any clinically significant chronic or acute medical condition that makes the volunteer unsuitable for participation
* History or evidence of drug or alcohol abuse
* History of intolerance to SC injection

Parts B/C MAD:

Inclusion Criteria:

* Male or female age 18 - 65
* BMI 18 - 32 kg/m^2
* Chronic HBV infection for >/= 6 months

Exclusion Criteria:

* Any clinically significant chronic or acute medical condition that makes the volunteer unsuitable for participation
* Significant fibrosis or cirrhosis
* History or evidence of drug or alcohol abuse
* History of intolerance to SC injection
* History of chronic liver disease from any cause other than chronic HBV infection
* History of hepatic decompensation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (3):
  - Investigative Site, Birtinya, Queensland
  - Investigative Site, Clayton, Victoria
  - Investigative Site, Fitzroy, Victoria
- Investigative Site, Hong Kong, Hong Kong
- Investigative Site, Auckland, New Zealand
- South Korea (2):
  - Investigative Site, Busan
  - Investigative Site, Seoul
- Thailand (3):
  - Investigative Site, Bangkok
  - Investigative Site, Hat Yai
  - Investigative Site, Khon Kaen

REFERENCES:
- [Derived] Yuen MF, Lim YS, Yoon KT, Lim TH, Heo J, Tangkijvanich P, Tak WY, Thanawala V, Cloutier D, Mao S, Arizpe A, Cathcart AL, Gupta SV, Hwang C, Gane E. VIR-2218 (elebsiran) plus pegylated interferon-alfa-2a in participants with chronic hepatitis B virus infection: a phase 2 study. Lancet Gastroenterol Hepatol. 2024 Dec;9(12):1121-1132. doi: 10.1016/S2468-1253(24)00237-1. Epub 2024 Oct 8. PMID 39389081
- [Derived] Gane E, Lim YS, Kim JB, Jadhav V, Shen L, Bakardjiev AI, Huang SA, Cathcart AL, Lempp FA, Janas MM, Cloutier DJ, Kaittanis C, Sepp-Lorenzino L, Hinkle G, Taubel J, Haslett P, Milstein S, Anglero-Rodriguez YI, Hebner CM, Pang PS, Yuen MF. Evaluation of RNAi therapeutics VIR-2218 and ALN-HBV for chronic hepatitis B: Results from randomized clinical trials. J Hepatol. 2023 Oct;79(4):924-932. doi: 10.1016/j.jhep.2023.05.023. Epub 2023 Jun 7. PMID 37290591
- [Derived] Gupta SV, Fanget MC, MacLauchlin C, Clausen VA, Li J, Cloutier D, Shen L, Robbie GJ, Mogalian E. Clinical and Preclinical Single-Dose Pharmacokinetics of VIR-2218, an RNAi Therapeutic Targeting HBV Infection. Drugs R D. 2021 Dec;21(4):455-465. doi: 10.1007/s40268-021-00369-w. Epub 2021 Nov 6. PMID 34741731

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A SAD VIR-2218 900 mg: Healthy subjects received a single dose of VIR-2218 of 900 mg administered SC
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part C: MAD 200 mg: Chronic HBV, HBeAg positive, subjects received 2 SC doses of 200 mg VIR-2218 administered 4 weeks apart.
  VIR-2218: VIR-2218 given by subcutaneous injection
Period: Overall Study
Arm/Group | Part A: SAD VIR-2218 50 mg | Part A: SAD VIR-2218 100 mg | Part A: SAD VIR-2218 200 mg | Part A: SAD VIR-2218 400 mg | Part A: SAD VIR-2218 600 mg | Part A SAD VIR-2218 900 mg | Part A: SAD Placebo | Part B: MAD VIR-2218 20 mg | Part B: MAD VIR-2218 50 mg | Part B: MAD VIR-2218 100 mg | Part B: MAD VIR-2218 200 mg | Part C: MAD VIR-2218 50 mg | Part C: MAD 200 mg | Part B: MAD Placebo | Part C: MAD Placebo
Started | 6 | 6 | 6 | 8 | 6 | 6 | 12 | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 2
Dosed | 6 | 6 | 6 | 7 (1 subject was not dosed and therefore not included in any analyses.) | 6 | 6 | 12 | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 2
Completed | 6 | 6 | 5 (1 Subject could not attend last follow up (Week 12 visit)) | 5 | 6 | 6 | 12 | 3 | 6 | 6 | 3 | 3 | 2 (1 non-treatment related SAE of suicide during follow up period) | 6 | 2
Not Completed | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Overall Number of Baseline Participants is not consistent with numbers provided in the rows of the Participant Flow module because we enrolled and randomized 8 participants for the Part A 400 mg cohort, but only 7 of these participants were dosed and included for full analysis dataset. We have added a row for dosed participants in the Participant Flow module, to clarify this inconsistency and reflect the number of participants in the analysis dataset.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: SAD VIR-2218 50 mg | Part A: SAD VIR-2218 100 mg | Part A: SAD VIR-2218 200 mg | Part A: SAD VIR-2218 400 mg | Part A: SAD VIR-2218 600 mg | Part A: SAD VIR-2218 900 mg | Part A: SAD Placebo | Part B: MAD VIR-2218 20 mg | Part B: MAD VIR-2218 50 mg | Part B: MAD VIR-2218 100 mg | Part B: MAD VIR-2218 200 mg | Part C: MAD VIR-2218 50 mg | Part C: MAD VIR-2218 200 mg | Part B: MAD Placebo | Part C: MAD Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 6 | 12 | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 2 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25 (3) | 23.3 (4) | 26.7 (3.8) | 24.3 (3.7) | 28.8 (6.3) | 32.5 (9.5) | 26.5 (6.7) | 40.3 (9.1) | 42.5 (10.8) | 45.2 (5.5) | 55 (4) | 35 (9.8) | 33.7 (13.1) | 44 (7.2) | 58.5 (7.8) | 33.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 3 | 7 | 3 | 3 | 5 | 1 | 1 | 1 | 3 | 2 | 1 | 3 | 1 | 44
  Male | 0 | 2 | 3 | 0 | 3 | 3 | 7 | 2 | 5 | 5 | 0 | 1 | 2 | 3 | 1 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 6 | 6 | 6 | 7 | 6 | 5 | 11 | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 2 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 0 | 0 | 2 | 1 | 1 | 3 | 5 | 5 | 3 | 3 | 3 | 6 | 2 | 39
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 5 | 5 | 3 | 3 | 8 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Region of Enrollment [Number; unit: participants]
  New Zealand | 6 | 6 | 6 | 7 | 6 | 6 | 12 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 54
  South Korea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 8
  Hong Kong | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 2 | 0 | 8
  Australia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 4
  Thailand | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 7
Hepatitis B Surface Antigen Levels (IU/mL) [Mean (Standard Deviation); unit: IU/mL] — HBsAg Levels seen across dose levels for Chronic Hepatitis B Subjects. Population: HBsAg levels would not be seen in Healthy subjects population, therefore 0 subjects were analyzed in corresponding dose levels.
  IU/mL
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 2 | 32
    (all) |  |  |  |  |  |  |  | 2372.227 (1168.940) | 3872.625 (5678.292) | 4009.863 (5239.703) | 2374.423 (2078.034) | 3488.037 (2454.215) | 12640.983 (10495.983) | 4819.127 (6348.594) | 1886.045 (1223.655) | 4456.52 (5657.74)
Alanine Aminotransferase Levels [Mean (Standard Deviation); unit: U/L] — Alanine Aminotransferase Levels in Chronic Hepatitis B Subjects Population: Alanine Aminotransferase Levels were not analyzed in Healthy subjects population.
  U/L
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 2 | 32
    (all) |  |  |  |  |  |  |  | 15.3 (4.6) | 23.5 (14.9) | 14.3 (5.0) | 10.0 (4.0) | 27.7 (18.6) | 26.0 (17.7) | 21.8 (17.6) | 26.5 (10.6) | 20.25 (13.08)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs)
Description: Number of Subjects with Adverse Events as assessed by CTCAE v5.0. In our planned analysis for this outcome measure, incidence is defined as the number of participants with treatment emergent AEs (TEAEs) in relation to the total number of participants in the cohort.
Time Frame: Up to 364 days
Population: The Overall Number of Participants Analyzed is not consistent with numbers provided in the rows of the Participant Flow module because we enrolled and randomized 8 participants for the Part A 400 mg cohort, but only 7 of these participants were dosed and included for full analysis dataset. We have added a row for dosed participants in the Participant Flow module, to clarify this inconsistency and reflect the number of participants in the analysis dataset.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: SAD VIR-2219 900 mg: Healthy subjects received a single dose of VIR-2218 of 900 mg administered SC
  VIR-2218: VIR-2218 given by subcutaneous injection
Arm/Group | Part A: SAD VIR-2218 50 mg | Part A: SAD VIR-2218 100 mg | Part A: SAD VIR-2218 200 mg | Part A: SAD VIR-2218 400 mg | Part A: SAD VIR-2218 600 mg | Part A: SAD VIR-2219 900 mg | Part A: SAD Placebo | Part B: MAD VIR-2218 20 mg | Part B: MAD VIR-2218 50 mg | Part B: MAD VIR-2218 100 mg | Part B: MAD VIR-2218 200 mg | Part C: MAD VIR-2218 50 mg | Part C: MAD VIR-2218 200 mg | Part B: MAD Placebo | Part C: MAD Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 6 | 12 | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 2
Participants | 4 | 3 | 4 | 5 | 3 | 3 | 6 | 0 | 2 | 5 | 2 | 2 | 2 | 1 | 1

2. Primary Outcome: Clinical Assessments Including But Not Limited to Laboratory Test Results
Description: Number of participants with clinically significant abnormalities in vital signs, electrocardiogram (ECG), and laboratory parameters graded by CTCAE v5.0.
Time Frame: Up to 336 days
Population: Number of participants analyzed is inclusive of clinically significant Vital Signs, ECGs, and Lab Findings. The Overall Number of Participants Analyzed is not consistent with numbers provided in the rows of the Participant Flow module. This inconsistency has been explained in the Analysis Population Description in our First Primary Outcome Measure as well.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: SAD VIR-2218 50 mg | Part A: SAD VIR-2218 100 mg | Part A: SAD VIR-2218 200 mg | Part A: SAD VIR-2218 400 mg | Part A: SAD VIR-2218 600 mg | Part A: SAD VIR-2218 900 mg | Part A: SAD Placebo | Part B: MAD VIR-2218 20 mg | Part B: MAD VIR-2218 50 mg | Part B: MAD VIR-2218 100 mg | Part B: MAD VIR-2218 200 mg | Part C: MAD VIR-2218 50 mg | Part C: MAD VIR-2218 200 mg | Part B: MAD Placebo | Part C: MAD Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 6 | 12 | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 2
Participants
  CTCAE v5.0 Lab Grade 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  CTCAE v5.0 Lab Grade 1 | 3 | 3 | 3 | 4 | 4 | 3 | 7 | 2 | 4 | 5 | 3 | 3 | 3 | 3 | 2
  CTCAE v5.0 Lab Grade 2 | 1 | 2 | 1 | 1 | 1 | 3 | 3 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0
  CTCAE v5.0 Lab Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CTCAE v5.0 Lab Grade 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinically Significant Vital Signs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinically Significant ECG | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Maximum Plasma Concentration (ng/mL)
Description: VIR-2218 and metabolite Maximum Concentration in Plasma
Time Frame: Part A: predose on Day 1 and at 30 min, 1h, 2h, 4h, 6h, 8h, 10h, 12h, 24h, 48h postdose and Week 1; Part B/C: predose on Day 1 and at 1h, 2h, 4h, 8h, 24h postdose, Week 1, predose on Week 4 and at 1h, 2h, 4h, 8h, 24h postdose, and Week 5
Population: The PK Analysis Set includes all randomized subjects who had at least 1 dose of VIR-2218 and 1 post-baseline PK parameter
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part B/C: MAD VIR-2218 20 mg: Chronic HBV subjects received 2 SC doses of 20 mg VIR-2218 administered 4 weeks apart.
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part B/C: MAD VIR-2218 50 mg: Chronic HBV subjects received 2 SC doses of 50 mg VIR-2218 administered 4 weeks apart.
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part B/C: MAD VIR-2218 100 mg: Chronic HBV, subjects received 2 SC doses of 100 mg VIR-2218 administered 4 weeks apart.
  VIR-2218: VIR-2218 given by subcutaneous injection
- Parts B/C: MAD VIR-2218 200 mg: Chronic HBV subjects received 2 SC doses of 200 mg VIR-2218 administered 4 weeks apart
  VIR-2218: VIR-2218 given by subcutaneous injection
Arm/Group | Part A: SAD VIR-2218 50 mg | Part A: SAD VIR-2218 100 mg | Part A: SAD VIR-2218 200 mg | Part A: SAD VIR-2218 400 mg | Part A: SAD VIR-2218 600 mg | Part A: SAD VIR-2218 900 mg | Part B/C: MAD VIR-2218 20 mg | Part B/C: MAD VIR-2218 50 mg | Part B/C: MAD VIR-2218 100 mg | Parts B/C: MAD VIR-2218 200 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 3 | 9 | 6 | 6
ng/mL
  VIR-2218 Cmax (Day 1): number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 2 | 7 | 6 | 6
  VIR-2218 Cmax (Day 1) | 155 (65.3) | 355 (117) | 711 (207) | 2110 (722) | 1830 (615) | 5010 (630) | 73.5 (NA) — SD is not reported when n<3. Not calculable; measurable in 2/3 subjects. | 118 (61.2) | 235 (79.0) | 826 (336)
  AS (N-1)3' VIR-2218 Cmax (Day 1): number analyzed (Participants) | 6 | 2 | 6 | 6 | 6 | 6 | 3 | 9 | 6 | 2
  AS (N-1)3' VIR-2218 Cmax (Day 1) | NA (NA) — Values were below the limit of quantification | 40.5 (NA) — SD is not reported when n<3 | 62.4 (17.6) | 259 (114) | 177 (99.2) | 514 (106) | NA (NA) — Values were below the limit of quantification | NA (NA) — Values were below the limit of quantification | NA (NA) — Values were below the limit of quantification | 66.1 (NA) — SD is not reported when n<3. Not calculable; measurable in 2/6 subjects.
  VIR-2218 Cmax (Day 29): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 8 | 6 | 6
  VIR-2218 Cmax (Day 29) |  |  |  |  |  |  | 51.8 (21.1) | 115 (38.2) | 256 (167) | 807 (374)
  AS (N-1)3' VIR-2218 Cmax (Day 29): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 9 | 1 | 3
  AS (N-1)3' VIR-2218 Cmax (Day 29) |  |  |  |  |  |  | NA (NA) — Values were below the limit of quantification | NA (NA) — Values were below the limit of quantification | NA (NA) — Mean not calculable if n=1 | 75.1 (27.2)

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (h)
Description: VIR-2218 and metabolite time of Cmax in Plasma: Median (Inter-Quartile Range Q1-Q3)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: h
Groups:
- Part B/C: MAD VIR-2218 20 mg: Chronic HBV, subjects received 2 SC doses of 20 mg VIR-2218 administered 4 weeks apart
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part B/C: MAD VIR-2218 100 mg: Chronic HBV subjects received 2 SC doses of 100 mg VIR-2218 administered 4 weeks apart.
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part B/C: MAD VIR-2218 200 mg: Chronic HBV, subjects received 2 SC doses of 200 mg VIR-2218 administered 4 weeks apart.
  VIR-2218: VIR-2218 given by subcutaneous injection
Arm/Group | Part A: SAD VIR-2218 50 mg | Part A: SAD VIR-2218 100 mg | Part A: SAD VIR-2218 200 mg | Part A: SAD VIR-2218 400 mg | Part A: SAD VIR-2218 600 mg | Part A: SAD VIR-2218 900 mg | Part B/C: MAD VIR-2218 20 mg | Part B/C: MAD VIR-2218 50 mg | Part B/C: MAD VIR-2218 100 mg | Part B/C: MAD VIR-2218 200 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 3 | 9 | 6 | 6
h
  VIR-2218 Tmax Day 1 | 4.25 [1.17 to 4.25] | 4.32 [4.25 to 6.17] | 5.21 [4.25 to 6.18] | 7.21 [4.25 to 8.25] | 7.21 [6.17 to 10.2] | 4.25 [4.25 to 8.25] | 4.00 [4.00 to 8.02] | 7.63 [4.00 to 7.93] | 2.48 [1.00 to 7.97] | 5.98 [3.98 to 8.00]
  AS(N-1)3' VIR-2218 Tmax Day 1: number analyzed (Participants) | 6 | 3 | 6 | 6 | 6 | 6 | 3 | 9 | 6 | 6
  AS(N-1)3' VIR-2218 Tmax Day 1 | NA [NA to NA] — Values were below the limit of quantification | 6.17 [4.25 to 6.17] | 6.17 [4.25 to 6.18] | 9.21 [4.25 to 10.2] | 10.2 [8.25 to 10.2] | 8.25 [4.25 to 10.2] | NA [NA to NA] — Values were below the limit of quantification | NA [NA to NA] — Values were below the limit of quantification | NA [NA to NA] — Values were below the limit of quantification | 8.00 [7.97 to 8.00]
  VIR-2218 Tmax Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 9 | 6 | 6
  VIR-2218 Tmax Day 29 |  |  |  |  |  |  | 3.95 [0.92 to 4.00] | 4.00 [4.00 to 7.98] | 8.00 [4.00 to 8.00] | 3.99 [2.00 to 8.00]
  AS (N-1)3' VIR-2218 Tmax Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 9 | 2 | 6
  AS (N-1)3' VIR-2218 Tmax Day 29 |  |  |  |  |  |  | NA [NA to NA] — Values were below the limit of quantification | NA [NA to NA] — Values were below the limit of quantification | 6.00 [4.00 to 8.00] | 5.99 [4.00 to 8.00]

5. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (ng*h/mL)
Description: VIR-2218 and metabolite Area under the curve from time 0 to last measurable Time
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Part B/C: MAD VIR-2218 20mg: Chronic HBV, subjects received 2 SC doses of 20 mg VIR-2218 administered 4 weeks apart
  VIR-2218: VIR-2218 given by subcutaneous injection
Arm/Group | Part A: SAD VIR-2218 50 mg | Part A: SAD VIR-2218 100 mg | Part A: SAD VIR-2218 200 mg | Part A: SAD VIR-2218 400 mg | Part A: SAD VIR-2218 600 mg | Part A: SAD VIR-2218 900 mg | Part B/C: MAD VIR-2218 20mg | Part B/C: MAD VIR-2218 50 mg | Part B/C: MAD VIR-2218 100 mg | Part B/C: MAD VIR-2218 200 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 3 | 9 | 6 | 6
h*ng/mL
  VIR-2218 AUClast (Day 1) | 1270 (270) | 3740 (1190) | 6630 (1160) | 23500 (2700) | 27900 (7540) | 58800 (9070) | 360 (199) | 1000 (285) | 2700 (943) | 9570 (2410)
  AS(N-1) 3' VIR-2218 AUClast (Day 1): number analyzed (Participants) | 6 | 3 | 6 | 6 | 6 | 6 | 3 | 9 | 6 | 6
  AS(N-1) 3' VIR-2218 AUClast (Day 1) | NA (NA) — Values were below the Limit of quantification | 208 (190) | 481 (149) | 2530 (613) | 2680 (1460) | 6430 (1500) | NA (NA) — Values were below the Limit of quantification | NA (NA) — Values were below the Limit of quantification | NA (NA) — Values were below the Limit of quantification | 482 (199)
  VIR-2218 AUClast (Day 29): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 9 | 6 | 6
  VIR-2218 AUClast (Day 29) |  |  |  |  |  |  | 339 (171) | 910 (326) | 2550 (638) | 9580 (3240)
  AS(N-1) 3' VIR-2218AUClast (Day 29): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 9 | 2 | 6
  AS(N-1) 3' VIR-2218AUClast (Day 29) |  |  |  |  |  |  | NA (NA) — Values were below the Limit of quantification | NA (NA) — Values were below the Limit of quantification | 174 (NA) — SD not calculated when n < 3 | 393 (230)

6. Secondary Outcome: Apparent Terminal Elimination Half-life (h)
Description: VIR-2218 Apparent Elimination Half-life t1/2 in Plasma: Median (Inter-Quartile Range Q1-Q3)
Time Frame: Part A: predose on Day 1 and at 30 min, 1h, 2h, 4h, 6h, 8h, 10h, 12h, 24h, 48h postdose and Week 1
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: h
Arm/Group | Part A: SAD VIR-2218 50 mg | Part A: SAD VIR-2218 100 mg | Part A: SAD VIR-2218 200 mg | Part A: SAD VIR-2218 400 mg | Part A: SAD VIR-2218 600 mg | Part A: SAD VIR-2218 900 mg
Number analyzed (Participants) | 5 | 4 | 5 | 6 | 6 | 6
h | 2.45 [2.35 to 3.26] | 3.64 [3.49 to 4.95] | 4.38 [4.22 to 6.11] | 3.54 [2.49 to 5.51] | 5.28 [5.12 to 5.62] | 4.55 [3.25 to 4.69]

7. Secondary Outcome: Apparent Plasma Clearance (L/h)
Description: VIR-2218 CL/F Apparent plasma clearance
Time Frame: Part A: predose on Day 1 and at 30 min, 1h, 2h, 4h, 6h, 8h, 10h, 12h, 24h, 48h postdose, and Week 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part A: SAD VIR-2218 50 mg | Part A: SAD VIR-2218 100 mg | Part A: SAD VIR-2218 200 mg | Part A: SAD VIR-2218 400 mg | Part A: SAD VIR-2218 600 mg | Part A: SAD VIR-2218 900 mg
Number analyzed (Participants) | 5 | 4 | 5 | 6 | 6 | 6
L/h | 34.0 (2.54) | 21.8 (4.27) | 30.8 (4.51) | 16.8 (1.76) | 21.9 (6.91) | 15.3 (2.08)

8. Secondary Outcome: Apparent Volume of Distribution (L)
Description: VIR-2218 VZ/F apparent volume of distribution
Time Frame: Part A: predose on Day 1 and at 30 min, 1h, 2h, 4h, 6h, 8h, 10h, 12h, 24h, 48h postdose, and Week 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Part A: SAD VIR-2218 50 mg | Part A: SAD VIR-2218 100 mg | Part A: SAD VIR-2218 200 mg | Part A: SAD VIR-2218 400 mg | Part A: SAD VIR-2218 600 mg | Part A: SAD VIR-2218 900 mg
Number analyzed (Participants) | 5 | 4 | 5 | 6 | 6 | 6
L | 155 (69.7) | 132 (40.7) | 223 (76.0) | 104 (62.6) | 176 (60.8) | 92.9 (24.6)

9. Secondary Outcome: Urine %fe 0-24h
Description: VIR-2218 and metabolite: Fraction excreted in the urine from time 0 to 24 h. Pooled Urine PK samples was collected at pre-specified intervals in the single ascending dose study of VIR-2218. Therefore, the following PK parameter, fraction excreted in the urine ( %fe 0-24h ) was only calculated in healthy subjects who participated in Part A of the study. This parameter was not listed as a secondary endpoint for parts B/C in the submitted protocol, and as such was not reported in this secondary outcome measures.
Time Frame: Pooled urine was collected at time interval D1 (0-4 hrs) (4-8 hrs) (8-12 hrs) and (12-24 hrs)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: % excreted in the urine from time 0-24h
Groups:
- Part A SAD: VIR-2218 50 mg: Healthy subjects received a single dose of VIR-2218 of 50 mg administered SC
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part A SAD: VIR-2218 100 mg: Healthy subjects received a single dose of VIR-2218 of 100 mg administered SC
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part A SAD: VIR-2218 200 mg: Healthy subjects received a single dose of VIR-2218 of 200 mg administered SC
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part A SAD: VIR-2218 400 mg: Healthy subjects received a single dose of VIR-2218 of 400 mg administered SC
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part A SAD: VIR-2218 600 mg: Healthy subjects received a single dose of VIR-2218 of 600 mg administered SC
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part A SAD: VIR-2218 900 mg: Healthy subjects received a single dose of VIR-2218 of 900 mg administered SC
  VIR-2218: VIR-2218 given by subcutaneous injection
Arm/Group | Part A SAD: VIR-2218 50 mg | Part A SAD: VIR-2218 100 mg | Part A SAD: VIR-2218 200 mg | Part A SAD: VIR-2218 400 mg | Part A SAD: VIR-2218 600 mg | Part A SAD: VIR-2218 900 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6
% excreted in the urine from time 0-24h
  VIR-2218 fe 0-24 | 16.9 (3.19) | 21.7 (6.22) | 23.2 (4.34) | 29.5 (5.72) | 32.3 (11.7) | 47.6 (8.59)
  AS(N-1)3' VIR-2218 fe 0-24 | 1.94 (0.480) | 4.16 (2.28) | 3.31 (0.656) | 4.99 (0.740) | 4.12 (2.31) | 6.96 (1.47)

10. Secondary Outcome: Apparent Renal Clearance (CLR/F)
Description: VIR-2218 Apparent renal clearance from 0 to 24 h. Pooled Urine PK samples was collected at pre-specified intervals in the single ascending dose study of VIR-2218. Therefore, the following PK parameter, apparent renal clearance (CLR/F) was only calculated in healthy subjects who participated in Part A of the study. This parameter was not listed as a secondary endpoint for parts B/C in the submitted protocol, and as such was not reported in this secondary outcome measures.
Time Frame: Pooled Urine was collected at time interval D1 (0-4 hrs) (4-8 hrs) (8-12 hrs) and (12-24 hrs)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part A: SAD VIR-2218 50 mg | Part A: SAD VIR-2218 100 mg | Part A: SAD VIR-2218 200 mg | Part A: SAD VIR-2218 400 mg | Part A: SAD VIR-2218 600 mg | Part A: SAD VIR-2218 900 mg
Number analyzed (Participants) | 5 | 4 | 5 | 6 | 6 | 6
L/h | 5.87 (0.728) | 5.22 (1.27) | 7.00 (0.659) | 5.13 (0.850) | 7.22 (1.480) | 7.47 (1.340)

11. Secondary Outcome: Maximum Reduction of Serum HBsAg From Baseline
Description: Maximum reduction of serum HBsAg from Day 1 until Week 16.
Time Frame: Up to 112 days
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Groups:
- Part B MAD: VIR-2218 20 mg: Chronic HBV, HBeAg negative, subjects received 2 SC doses of 20 mg VIR-2218 administered 4 weeks apart
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part B MAD: VIR-2218 50 mg: Chronic HBV, HBeAg negative, subjects received 2 SC doses of 50 mg VIR-2218 administered 4 weeks apart
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part B MAD: VIR-2218 100 mg: Chronic HBV, HBeAg negative, subjects received 2 SC doses of 100 mg VIR-2218 administered 4 weeks apart
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part B MAD: VIR-2218 200 mg: Chronic HBV, HBeAg negative, subjects received 2 SC doses of 200 mg VIR-2218 administered 4 weeks apart
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part C MAD: VIR-2218 50 mg: Chronic HBV, HBeAg positive, subjects received 2 SC doses of 50 mg VIR-2218 administered 4 weeks apart
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part C MAD: VIR-2218 200 mg: Chronic HBV, HBeAg positive, subjects received 2 SC doses of 200 mg VIR-2218 administered 4 weeks apart
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part B MAD: Placebo: Chronic HBV, HBeAg negative, subjects received 2 SC doses of placebo administered 4 weeks apart
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part C MAD: Placebo: Chronic HBV, HBeAg positive, subjects received 2 SC doses of placebo administered 4 weeks apart
  VIR-2218: VIR-2218 given by subcutaneous injection
Arm/Group | Part B MAD: VIR-2218 20 mg | Part B MAD: VIR-2218 50 mg | Part B MAD: VIR-2218 100 mg | Part B MAD: VIR-2218 200 mg | Part C MAD: VIR-2218 50 mg | Part C MAD: VIR-2218 200 mg | Part B MAD: Placebo | Part C MAD: Placebo
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 2
log10 IU/mL | -1.031 (0.574) | -1.230 (0.702) | -1.504 (0.540) | -1.653 (0.154) | -1.161 (0.350) | -1.568 (0.636) | -0.098 (0.047) | -0.068 (0.01)

12. Secondary Outcome: Number of Subjects With Serum HBsAg Loss at Any Time Point
Description: Serum HBsAg loss is defined as quantitative HBsAg < 0.05 IU/mL at two or more consecutive measurements
Time Frame: Up to 336 days
Measure: Count of Participants; unit: Participants
Groups:
- Part B MAD: VIR-2218 50 mg: Chronic HBV, HBeAg negative, subjects received 2 SC doses of 50 mg VIR-2218 administered 4 weeks apart.
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part B MAD: VIR-2218 100 mg: Chronic HBV, HBeAg negative, subjects received 2 SC doses of 100 mg VIR-2218 administered 4 weeks apart.
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part B MAD: VIR-2218 200 mg: Chronic HBV, HBeAg negative, subjects received 2 SC doses of 200 mg VIR-2218 administered 4 weeks apart.
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part C MAD: VIR-2218 50 mg: Chronic HBV, HBeAg positive, subjects received 2 SC doses of 50 mg VIR-2218 administered 4 weeks apart.
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part C MAD: VIR-2218 200 mg: Chronic HBV, HBeAg positive, subjects received 2 SC doses of 200 mg VIR-2218 administered 4 weeks apart.
  VIR-2218: VIR-2218 given by subcutaneous injection
- Part B MAD: Placebo: Chronic HBV, HBeAg negative, subjects received 2 SC doses of placebo administered 4 weeks apart.
  Placebo: Sterile normal saline (0.9% NaCl) given by subcutaneous injection
- Part C MAD: Placebo: Chronic HBV, HBeAg positive, subjects received 2 SC doses of placebo administered 4 weeks apart.
  Placebo: Sterile normal saline (0.9% NaCl) given by subcutaneous injection
Arm/Group | Part B MAD: VIR-2218 20 mg | Part B MAD: VIR-2218 50 mg | Part B MAD: VIR-2218 100 mg | Part B MAD: VIR-2218 200 mg | Part C MAD: VIR-2218 50 mg | Part C MAD: VIR-2218 200 mg | Part B MAD: Placebo | Part C MAD: Placebo
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Subjects With Sustained Serum HBsAg Loss for >/= 6 Months
Description: Serum HBsAg loss is defined as quantitative HBsAg < 0.05 IU/mL at two or more consecutive measurements
Time Frame: Up to 336 days
Measure: Count of Participants; unit: Participants
Arm/Group | Part B MAD: VIR-2218 20 mg | Part B MAD: VIR-2218 50 mg | Part B MAD: VIR-2218 100 mg | Part B MAD: VIR-2218 200 mg | Part C MAD: VIR-2218 50 mg | Part C MAD: VIR-2218 200 mg | Part B MAD: Placebo | Part C MAD: Placebo
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Subjects With Anti-HBs Seroconversion at Any Timepoint
Description: Anti-HBs seroconversion is defined as anti-HBs positivity at two or more consecutive measurements
Time Frame: Up to 336 days
Measure: Count of Participants; unit: Participants
Groups:
- Part B MAD: VIR-2218 20 mg: Chronic HBV, HBeAg negative, subjects received 2 SC doses of 20 mg VIR-2218 administered 4 weeks apart.
  VIR-2218: VIR-2218 given by subcutaneous injection
Arm/Group | Part B MAD: VIR-2218 20 mg | Part B MAD: VIR-2218 50 mg | Part B MAD: VIR-2218 100 mg | Part B MAD: VIR-2218 200 mg | Part C MAD: VIR-2218 50 mg | Part C MAD: VIR-2218 200 mg | Part B MAD: Placebo | Part C MAD: Placebo
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Subjects With HBeAg Loss and/or Anti-HBe Seroconversion at Any Timepoint
Description: HBeAg loss is defined as quantitative HBeAg < 0.11 IU/mL at two or more consecutive measurements. anti-HBe seroconversion is defined as anti-HBe positivity at two or more consecutive measurements
Time Frame: Up to 336 days
Measure: Count of Participants; unit: Participants
Arm/Group | Part C MAD: VIR-2218 50 mg | Part C MAD: VIR-2218 200 mg | Part C MAD: Placebo
Number analyzed (Participants) | 3 | 3 | 2
Participants
  Number of Subjects with HBeAg Loss | 0 | 1 | 0
  Number of Subjects with anti-HBe seroconversion | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 364 days after first dose with VIR-2218 or placebo
Description: The Total Number of Participants at Risk - All Cause Mortality, Serious Adverse Events, and Other (Not Including Adverse Events) tables - is not consistent with numbers provided in the rows of the Participant Flow module. This inconsistency has been explained in the Baseline Analysis Population Description.
Groups:
- Part A SAD: Placebo: Healthy subjects received a single dose of placebo administered SC
  Placebo: Sterile normal saline (0.9% NaCl) given by subcutaneous injection
Arm/Group | Part A SAD: VIR-2218 50 mg | Part A SAD: VIR-2218 100 mg | Part A SAD: VIR-2218 200 mg | Part A SAD: VIR-2218 400 mg | Part A SAD: VIR-2218 600 mg | Part A SAD: VIR-2218 900 mg | Part A SAD: Placebo | Part B MAD: VIR-2218 20 mg | Part B MAD: VIR-2218 50 mg | Part B MAD: VIR-2218 100 mg | Part B MAD: VIR-2218 200 mg | Part C MAD: VIR-2218 50 mg | Part C MAD: VIR-2218 200 mg | Part B MAD: Placebo | Part C MAD: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/12 | 0/3 | 0/6 | 0/6 | 0/3 | 0/3 | 1/3 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/12 | 0/3 | 0/6 | 1/6 | 0/3 | 0/3 | 0/3 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 4/6 | 3/6 | 4/6 | 5/7 | 3/6 | 3/6 | 6/12 | 0/3 | 2/6 | 5/6 | 2/3 | 2/3 | 2/3 | 1/6 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A SAD: VIR-2218 50 mg (N=6) | Part A SAD: VIR-2218 100 mg (N=6) | Part A SAD: VIR-2218 200 mg (N=6) | Part A SAD: VIR-2218 400 mg (N=7) | Part A SAD: VIR-2218 600 mg (N=6) | Part A SAD: VIR-2218 900 mg (N=6) | Part A SAD: Placebo (N=12) | Part B MAD: VIR-2218 20 mg (N=3) | Part B MAD: VIR-2218 50 mg (N=6) | Part B MAD: VIR-2218 100 mg (N=6) | Part B MAD: VIR-2218 200 mg (N=3) | Part C MAD: VIR-2218 50 mg (N=3) | Part C MAD: VIR-2218 200 mg (N=3) | Part B MAD: Placebo (N=6) | Part C MAD: Placebo (N=2)
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A SAD: VIR-2218 50 mg (N=6) | Part A SAD: VIR-2218 100 mg (N=6) | Part A SAD: VIR-2218 200 mg (N=6) | Part A SAD: VIR-2218 400 mg (N=7) | Part A SAD: VIR-2218 600 mg (N=6) | Part A SAD: VIR-2218 900 mg (N=6) | Part A SAD: Placebo (N=12) | Part B MAD: VIR-2218 20 mg (N=3) | Part B MAD: VIR-2218 50 mg (N=6) | Part B MAD: VIR-2218 100 mg (N=6) | Part B MAD: VIR-2218 200 mg (N=3) | Part C MAD: VIR-2218 50 mg (N=3) | Part C MAD: VIR-2218 200 mg (N=3) | Part B MAD: Placebo (N=6) | Part C MAD: Placebo (N=2)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 2 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may discuss or publish results after:

* the study results in their entirety have been publicly disclosed by or with the consent of the Sponsor OR study has been completed at all investigative sites for at least 2 years
* provision of publication up to 60 days before planned submission to allow Sponsor to remove confidential information or identify Sponsor intellectual property

Publication may be delayed as applicable, up to 120 days for Sponsor to file patent application(s)

DOCUMENTS (2):
  • Study Protocol (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/88/NCT03672188/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT03672188/SAP_001.pdf